CLINICAL TRIAL: NCT07228702
Title: Bacteriophage Therapy for Mycobacterium Abscessus Pulmonary Infection: An Open Label Individual Patient Study
Brief Title: Bacteriophage Therapy for Mycobacterium Abscessus Pulmonary Infection
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Vancouver Coastal Health (Other Government)
Responsible Party: Principal Investigator, William Connors, Clinical Associate Professor, Vancouver Coastal Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPHAGE-2025-01; Control # 300143 (Other: Health Canada)
Record Dates: First submitted 2025-09-09; First posted 2025-11-14 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Non-Tuberculous Mycobacterial (NTM) Pneumonia; Mycobacterium Abscessus Infection
Keywords: non-tuberculous mycobacteria; bacteriophage; mycobacteriophage; mycobacterium abscessus; pulmonary disease
MeSH Terms: conditions — Pneumonia; Mycobacterium Infections, Nontuberculous; Lung Diseases | interventions — Amikacin; Clofazimine; bedaquiline; Linezolid; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Use of mycobacteriophage
  Interventions: Biological: Mycobacteriophage Muddy_HRMN0052; Drug: Amikacin Injection; Drug: Clofazimine; Drug: Bedaquiline (B); Drug: Linezolid (LZD); Drug: Sulfamethoxazole/Trimethoprim

INTERVENTIONS:
Biological: Mycobacteriophage Muddy_HRMN0052 — In-vitro effective Mycobacteriophage Muddy_HRMN0052 against specific strain of Mycobacterium abscessus ssp abscessuss
Drug: Amikacin Injection — Amikacin 1000mg IV 3x/wk
Drug: Clofazimine — Clofazimine 100mg PO OD
Drug: Bedaquiline (B) — Bedaquiline 400mg PO OD x 2 weeks then 200mg PO 3x/wk (Alternate agent if toxicity/intolerance to amikacin or clofazimine to ensure on 2 antibiotics throughout)
Drug: Linezolid (LZD) — Linezolid 600mg PO OD (dose reduce to 600mg PO 3x/wk if adverse effects)(Alternate agent if toxicity/intolerance to amikacin or clofazimine to ensure on 2 antibiotics throughout)
Drug: Sulfamethoxazole/Trimethoprim — Sulfamethoxazole/Trimethoprim 800/160mg PO BID (Alternate agent if toxicity/intolerance to amikacin or clofazimine to ensure on 2 antibiotics throughout)

SUMMARY:
This study aims to use mycobacteriophage therapy, using identified in-vitro effective Mycobacteriophage Muddy_HRMN0052, along with combination conventional antimycobacterial therapy for their NTM pulmonary disease with Mycobacterium abscessus with goal to reduce infection burden and improve pulmonary disease

DETAILED DESCRIPTION:
Hypothesis

Hypothesis: Mycobacteriophage therapy, using identified in-vitro effective Mycobacteriophage Muddy_HRMN0052, along with combination conventional antimycobacterial therapy for their NTM pulmonary disease with MABS will reduce infection burden and improve pulmonary disease.

Objectives:

1. Efficacy - Assess MABS pulmonary disease response mycobacteriophage therapy
2. Safety - Determine tolerability and off target effects of IV and inhaled mycobacteriophage therapy

Specific End Points (during and post treatment up to last clinical follow-up (>24month):

1. Microbiologic: Time to sputum smear and culture conversion; durability of sputum culture conversion during and post treatment; change in sputum microbiology on and post treatment; change in MABS drug and mycobacteriophage susceptibility on and post treatment; mycobacteriophage neutralizing antibody development.
2. Clinical: Pulmonary and systemic symptom report; sputum production volume (patient report); chest imaging response (CT scan); Spirometry and full PFT; quality of life
3. Other: Adverse clinical and laboratory events

Information on the Investigational Product (Mycobacteriophage Muddy_HRMN0052):

1. Mechanism of action Bacteriophage therapy (phage therapy) involves the use of live, lytic bacteriophages to treat bacterial infections via bacterial cell lysis. Lytic bacteriophages mediate their antimicrobial effect by way of specific attachment to bacterial cell wall receptors, injection of bacteriophage DNA into the bacterium, recruitment of bacterial host cell machinery for bacteriophage protein production, and subsequent lysis of the bacterial cell with release of bacteriophage progeny.
2. Dose, frequency, route of administration for the product

Initial IV dosing of Mycobacteriophage Muddy_HRMN0052 for treatment of Mycobacterium abscessus should be 1mL containing 1 x 10^9 PFU/mL to be given IV twice daily.

Inhalation:

Initial inhaled (by nebulization or aerosolization) dosing of Mycobacteriophage Muddy_HRMN0052 for treatment of Mycobacterium abscessus should be 1mL containing 1 x 10^9 PFU/mL to be given inhaled twice daily. For inhaled use, Mycobacteriophage Muddy_HRMN0052 is supplied in the lyophilized form that enhances the stability during nebulization.

The treatment duration for both routes of administration is expected to be between 16 to 24 weeks at minimum with a possible extension up to 24 months if necessary, based upon clinical response.

Treatment Regimen and Duration:

Initial IV dosing for treatment of Mycobacterium abscessus with Mycobacteriophage Muddy_HRMN0052 should be 1mL containing 1 x 10^9 PFU/mL to be given IV twice daily.

Initial inhaled dosing for treatment of Mycobacterium abscessus with Mycobacteriophage Muddy_HRMN0052 should be 1mL containing 1 x 10^9 PFU/mL to be given inhaled twice daily.

The duration of treatment to be determined based on clinical response, but the recommended initial course of treatment is expected to be at least 16-24 weeks and used together with antimicrobial therapy targeted at the infecting organism recovered from the patient. The duration and start timing of IV and inhaled formulation will be guided by tolerance and clinical response with potential transition to single route as treatment progresses.

If the inhaled route of administration is not tolerated by the patient, as determined by a drop in FEV1 percent predicted (FEV1pp) of greater than 20% from baseline with the first dosage, and/or intolerable symptoms of cough or shortness of breath that are not relieved with bronchodilator (salbutamol) with the first dose, or if respiratory symptoms develop with later dosing that are deemed intolerable by the patient, then the treatment will revert to IV administration.

Concurrent with MUDDY phage treatment the following antibiotics will be use. Use of phage plus antibiotics is similar to prior reported human treatment of NTM disease with mycobacteriophages and in line with Antibacterial Resistance Leadership Group (ARLG) Phage Taskforce (U.S.) guidance. To balance effectiveness and toxicity risk two antibiotics that Mycobacterium abscessus has been demonstrated susceptible to will be used. Selection of drugs is also informed by tolerance during prior treatment. Alternate medications will be used if toxicity from first choice antibiotics encountered. Antibiotics/rationale are as follows, all doses are standard weight-based dosing:

Initial Regimen:

1. Amikacin 1000mg IV 3x/wk - prior good tolerance, evidence based preferred agent for treatment of NTM disease
2. Clofazimine 100mg PO OD - prior good tolerance; general low toxicity profile, M. abscessus demonstrated to have favorable low MIC.

Alternate agents (use if toxicity/intolerance to initial regimen agents to ensure on 2 antibiotics throughout):

1. Bedaquiline 400mg PO OD x 2 weeks then 200mg PO 3x/wk - prior good tolerance; general low toxicity profile, M. abscessus demonstrated to have favorable low MIC.
2. Linezolid 600mg PO OD (dose reduce to 600mg PO 3x/wk if adverse effects) - unclear if contributed to prior anorexia while on multidrug regimen, risk of toxicity with extended use
3. Sulfamethoxazole/Trimethoprim 800/160mg PO BID - less evidence available supporting use for M. abscessus disease, prior issues with associated hyperkalemia

ELIGIBILITY:
This is an individual patient expanded access study specific to one individual based on tailor intervention (Mycobacteriophage)

Inclusion Criteria:

* consent to participation

Exclusion Criteria:

* non-consent to participation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Microbiologic: Response | 2 years
  1. Sputum culture status: time (days) to durable sputum culture conversion (no mycobacterial growth on 3 sputum sample)

SECONDARY OUTCOMES:
Microbiologic: Resistance development | 2 years
  MABS drug and phage resistance development on follow-up sputum cultures (on treatment and post)
Microbiologic: Neutralizing antibody status. | 2 years
  Detection of mycobacteriophage neutralizing antibodies on follow-up serology
Clinical: Symptoms | 2 year
  Pulmonary and systemic symptom report change using adapted global assessment of quality of life. This will be patient reported and scored at each clinical assessment as follows and in reference/comparison to last/most recent score (negative = worse, positive = improved):
  * 4 Markedly Improved ( >75% improved quality of life)
  * 3 Much Improved (51-75% improved quality of life)
  * 2 Improved (25-50% improved quality of life)
  * 1 Slightly Improved (1-24% improved quality of life) 0 No Change
    * 1 Slightly Worse (1-24% reduced quality of life)
    * 2 Worse (25-50% reduced quality of life)
    * 3 Much Worse (51-75% reduced quality of life)
    * 4 Markedly Worse (>75 % reduced quality of life)
Clinical: Sputum | 2 year
  sputum production volume change (patient report)
Clinical: Radiographic | 2 year
  Chest imaging response (CT scan) to treatment
Clinical: Pulmonary Function | 2 year
  Spirometry and full PFT changes on treatment
Clinical: Adverse effects | 2 year
  Adverse clinical and laboratory events (number and severity) on treatment
Clinical: Symptoms | 2 year
  Pulmonary and systemic symptom report change (Physicians Global Assessment to measure quality of life)

CONTACTS AND LOCATIONS:
Locations (1):
- Vancouver General Hospital Non-Tuberculous Mycobacterial Disease Clinic, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Will depend on participant and institution agreement

REFERENCES:
- [Background] Reindel R, Fiore CR. Phage Therapy: Considerations and Challenges for Development. Clin Infect Dis. 2017 Jun 1;64(11):1589-1590. doi: 10.1093/cid/cix188. No abstract available. PMID 28329182
- [Background] Hatfull GF. Phage Therapy for Nontuberculous Mycobacteria: Challenges and Opportunities. Pulm Ther. 2023 Mar;9(1):91-107. doi: 10.1007/s41030-022-00210-y. Epub 2022 Dec 30. PMID 36583829
- [Background] Dedrick RM, Smith BE, Cristinziano M, Freeman KG, Jacobs-Sera D, Belessis Y, Whitney Brown A, Cohen KA, Davidson RM, van Duin D, Gainey A, Garcia CB, Robert George CR, Haidar G, Ip W, Iredell J, Khatami A, Little JS, Malmivaara K, McMullan BJ, Michalik DE, Moscatelli A, Nick JA, Tupayachi Ortiz MG, Polenakovik HM, Robinson PD, Skurnik M, Solomon DA, Soothill J, Spencer H, Wark P, Worth A, Schooley RT, Benson CA, Hatfull GF. Phage Therapy of Mycobacterium Infections: Compassionate Use of Phages in 20 Patients With Drug-Resistant Mycobacterial Disease. Clin Infect Dis. 2023 Jan 6;76(1):103-112. doi: 10.1093/cid/ciac453. PMID 35676823